CLINICAL TRIAL: NCT04388488
Title: Connect TF - An Investigation of Function and Usability of a New Adaptable Socket System for
Brief Title: Connect TF - An Investigation of Function and Usability of a New Adaptable Socket System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP2020021338
Record Dates: First submitted 2020-04-30; First posted 2020-05-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Prosthesis User; Amputation

STUDY DESIGN:
Intervention Model Description: This clinical investigation will be of a single group non-randomized open label prospective repeated measures (ABBA) design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CONNECT TF (Experimental): Trans-femoral amputees currently using a conventional handmade socket will be fitted with the CONNECT TF adaptable socket system for 6 weeks and their current existing conventional socket for 6 weeks, data collection on both sockets will be performed and outcomes compared.
  Interventions: Device: CONNECT TF adaptable socket system; Device: Any conventional handmade socket

INTERVENTIONS:
Device: CONNECT TF adaptable socket system — Prefabricated, adaptable socket system
Device: Any conventional handmade socket — Subjects current socket

SUMMARY:
The primary objective of this investigation is to evaluate how the CONNECT TF compares to traditional handmade sockets, specifically that it provides reliable suspension and improved usability and comfort for the amputee, and that it enables single clinical visit for fitting.

DETAILED DESCRIPTION:
Design:

This clinical investigation will be of a single group non-randomized open label prospective repeated measures (ABBA) design comparing subject´s current conventional socket and the CONNECT TF. The subjects will be asked to use the CONNECT TF as their primary prosthesis for up to six weeks. Subject will be fitted with the same foot-pylon-knee prosthetic system as used with their current conventional socket, with the CONNECT TF socket.

Procedures:

There are four scheduled study events. At the initial visit, the first study event, for each subject a qualified researcher will obtain an informed consent. Prior to fitting the patient subject to CONNECT TF he/she will be asked to provide feedback and perform tasks on/using their current conventional prosthetic socket. The patient subjects will be fitted with the CONNECT TF within the standard methods of prosthetic fitting, alignment, introduction, training and walking on various terrain.

The CPO (Certified Prosthetis/Orthotist) will conduct the fitting and aligning of the CONNECT TF.

A Co-Investigator will time the fitting procedure; from unpacking the device until it is correctly adjusted and properly fit to the subject.

Data on initial feedback on the device will be collected from the subjects using the instruments specified above. Afterwards an appointment at 2 weeks is made and the subjects leave the clinic on the device.

If the fitting of CONNECT TF fails, i.e. the PI/CPO does not manage to fit the device properly or the subject cannot use the device as intended during training at the clinic, a new appointment is made, if the subject is willing to continue participation.

The second event will be according to the appointment scheduled 2 weeks earlier. During this visit the same set of information will be gathered from/on the subjects as at the initial visit using the conventional socket. A 6 week follow up (6WFU) visit is scheduled and the subject leaves on the CONNECT TF socket.

The third event will be according to the appointment scheduled at the previous visit. During this visit set of information will be gathered from/on the subjects as at the initial visit using the conventional socket. A final 6WFU visit is scheduled and the subjects are fitted back to and leave on their current conventional socket.

The fourth event will be according to the appointment scheduled at the previous visit. During this visit set of information will be gathered from/on the subjects as at the initial visit using the conventional socket. End of study.

Data analysis:

The dataset will be assessed with inferential statistics based on the acceptance criteria for the data, as applicable.

Outcomes at each time point will be visually inspected for normality using histograms and qq-plots. If the data are deemed to be normal the hypothesis will be tested using a two-tailed, paired, student's t-test for 2WFU evaluation and mixed models for the 6WFU evaluation. Non-normal data will be tested using the Wilcoxon signed-rank test.

ELIGIBILITY:
Inclusion Criteria:

* Lower limb amputees
* Uni- or bilateral TF amputees
* 40 < body weight < 125Kg
* Activity level: K1-K2;
* Liner size: 28-45;
* Max 1 user in sizes 28 and 45, respectively
* Residual limb parameters; perineum to distal end: 205 to 280 mm
* Older than 18 years
* Prosthetic users for more than 3 months
* Components of conventional socket functionally compatible to Össur components (foot-pylon-knee combination)
* Users understanding the function of the device
* Willing and able to participate in the study and follow the protocol

Exclusion Criteria:

* Other amputees
* 40> body weight > 125Kg
* Amputees with broken skin on the residual limb
* Younger than 18 years
* Prosthetic users for less than 3 months
* Using no liner
* Using a microprocessor controlled prosthetic knee not manufactured by Össur
* Users not understanding the function of the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Comprehensive Lower-limb Amputee Socket Survey (CLASS) | 6 weeks
  CLASS is a self-report measure of prosthetic socket satisfaction for lower limb amputees, designed to provide an effective means of communication for the patient to describe with clarity, the quality of their socket fit during common activities. CLASS evaluates static and dynamic features of socket stability, suspension, comfort and appearance and has been reported to be a reliable, quick and easy report measure.

SECONDARY OUTCOMES:
Prosthesis evaluation questionnaire - Residual limb health (PEQ- RLH) | 6 weeks
  average of 6 item subscale from the PEQ
Prosthesis evaluation questionnaire - Sounds (PEQ-Sounds) | 6 weeks
  average of 2 item subscale from the PEQ
Mobility (2MWT) | 6 weeks
  2 minute walking test
Balance during ambulation (TUG) | 6 weeks
  Times up and go test

CONTACTS AND LOCATIONS:
Overall Officials: Sashwati Roy, PhD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - IU Health Comprehensive Wound Center at Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No